CLINICAL TRIAL: NCT01466153
Title: A Phase 2 Open-label Study of MEDI-551 and Bendamustine vs Rituximab and Bendamustine in Adults With Relapsed or Refractory CLL
Brief Title: A Phase 2, Multicenter, Open-label Study of MEDI-551 in Adults With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-551-1019
Record Dates: First submitted 2011-09-30; First posted 2011-11-07 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic lymphocytic leukemia; leukemia; B-Cell malignancy; anti-CD19; monoclonal antibody; CLL; Refractory; Relapse; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Recurrence; Lymphoma, Non-Hodgkin | interventions — Rituximab; Bendamustine Hydrochloride; inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rituximab + Bendamustine (Active Comparator): Rituximab was administered by IV infusion as 375 mg/m^2 on Day 2 of Cycle 1 and then 500 mg/m^2 on Day 1 of up to 5 subsequent 28-day cycle. Bendamustine was also administered by IV infusion on Day 1 and Day 2 of every cycle (total 6 cycles). Bendamustine was administered before the administration of rituximab in each cycle.
  Interventions: Drug: Rituximab; Drug: Bendamustine
- MEDI-551 2 mg/kg + Bendamustine (Experimental): MEDI-551 2 mg/kg was administered by IV infusion on Days 2 and 8 of Cycle 1 and then on Day 1 of up to 5 subsequent 28-day cycle. Bendamustine was also administered by IV infusion on Day 1 and Day 2 of every cycle (total 6 cycles). Bendamustine was administered before the administration of MEDI-551 in each cycle.
  Interventions: Drug: Bendamustine; Drug: MEDI-551
- MEDI-551 4 mg/kg + Bendamustine (Experimental): MEDI-551 4 mg/kg was administered by IV infusion on Days 2 and 8 of Cycle 1 and then on Day 1 of up to 5 subsequent 28-day cycle. Bendamustine was also administered by IV infusion on Day 1 and Day 2 of every cycle (total 6 cycles). Bendamustine was administered before the administration of MEDI-551 in each cycle.
  Interventions: Drug: Bendamustine; Drug: MEDI-551

INTERVENTIONS:
Drug: Rituximab — Rituximab was administered by IV infusion as a dose of 375 mg/m^2 on Day 2 of Cycle 1 and then at 500 mg/m^2 on Day 1 of up to 5 subsequent 28-day cycles
  Other Names: Rituxan; MabThera
  Arms: Rituximab + Bendamustine
Drug: Bendamustine — Bendamustine was administered by IV infusion as a dose of 70 mg/m^2 on Day 1 and Day 2 of each 5 subsequent 28-day cycle.
Drug: MEDI-551 — MEDI-551 was administered at 2 mg/kg or 4 mg/kg by IV infusion on Days 2 and 8 of Cycle 1 and then on Day 1 of up to 5 subsequent 28-day cycles.
  Arms: MEDI-551 2 mg/kg + Bendamustine; MEDI-551 4 mg/kg + Bendamustine

SUMMARY:
The overall purpose of the study was to determine if MEDI-551, when used in combination with salvage chemotherapy (bendamustine) in participants with relapsed or refractory CLL who are not eligible for Autologous Stem Cell Transplant (ASCT), had superior efficacy compared to rituximab in the same population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell Chronic Lymphocytic Leukemia (CLL) according to the National Cancer Institute criteria; Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2; Adequate hematological function

Exclusion Criteria:

* Any chemotherapy, radiotherapy, immunotherapy, biologic, investigational, or hormonal therapy for treatment of lymphoma within 28 days prior to treatment;
* Exposure to bendamustine within the 180 days before study enrollment
* Prior autologous or allogeneic stem cell transplantation (SCT);
* Clinically significant abnormality on electrocardiogram (ECG) as determined by the treating physician or medical monitor;
* History of other invasive malignancy within 5 years except for localized/in situ carcinomas;
* Evidence of active infection, Confirmed current central nervous system involvement by leukemia or lymphoma;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-02-07; Primary Completion 2016-01-08 (Actual); Study Completion 2016-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, Study Director — MedImmune LLC
Locations (54):
- United States (14):
  - Research Site, Birmingham, Alabama
  - Research Site, Burbank, California
  - Research Site, La Jolla, California
  - Research Site, Palm Springs, California
  - Research Site, Skokie, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Fargo, North Dakota
  - Research Site, Dayton, Ohio
  - Research Site, Newark, Ohio
  - Research Site, Watertown, South Dakota
  - Research Site, Lubbock, Texas
  - Research Site, Morgantown, West Virginia
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Arlon
  - Research Site, Kortrijk
  - Research Site, Mons
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Canada (3):
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- France (7):
  - Research Site, Amiens
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Le Mans
  - Research Site, Libourne
  - Research Site, Marseille
  - Research Site, Nîmes
- Germany (5):
  - Research Site, Dortmund
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, München
  - Research Site, Würzburg
- Israel (2):
  - Research Site, Haifa
  - Research Site, Ramat Gan
- Italy (15):
  - Research Site, Bari
  - Research Site, Lecce
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Torino
  - Research Site, Udine
- Poland (2):
  - Research Site, Gdynia
  - Research Site, Warsaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 182 participants were screened and 159 participants were randomized.
Period: Overall Study
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Started | 62 | 36 | 61
Completed | 33 | 12 | 36
Not Completed | 29 | 24 | 25
Not completed — Disease Progression | 2 | 2 | 0
Not completed — Adverse Event | 14 | 13 | 17
Not completed — Withdrawal of Consent | 2 | 0 | 0
Not completed — Investigator Discretion | 3 | 2 | 2
Not completed — Randomized-Not Treated | 2 | 3 | 4
Not completed — Other-Unspecified | 6 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population includes all participants who were randomized into the study.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine | TOTAL
Number analyzed (Participants) | 62 | 36 | 61 | 159
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.4 (8.8) | 65.1 (8.7) | 66.3 (8.9) | 65.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 18 | 48
  Male | 46 | 22 | 43 | 111

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR, defined as the proportion of participants with complete response (CR) or partial response (PR) out of total number of participants. Responses were assessed by using National Cancer Institute - Working Group guidelines on CLL.
Time Frame: From treatment administration (Day 1) until disease progression, death, initiation of alternative therapy, withdrawal of consent, or end of study (up to 24 months)
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Percentage of Participants | 59.7 [46.4 to 71.9] | 52.8 [35.5 to 69.6] | 63.9 [50.6 to 75.8]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs MEDI-551 4 mg/kg + Bendamustine; Test type: Superiority or Other; p = 0.4475, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs) and Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug (MEDI-551). A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and Day 90 that were absent before treatment or that worsened relative to pre-treatment state. An AESIs was one of scientific and medical interest specific to understanding of study product and may have required close monitoring and rapid communication by investigator to the sponsor. Treatment emergent AESIs were collected from the time of dosing through Day 90 after the last dose of study drug.Hepatic function abnormality and infusion reactions resulting in discontinuation were considered as AESIs.
Time Frame: From time of consent to 90 days post last dose
Population: The safety population includes all participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 60 | 33 | 57
Participants
  TEAEs | 58 | 33 | 57
  TESAEs | 19 | 16 | 19
  AESIs | 2 | 4 | 6

3. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as AEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Laboratory evaluations (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: From time of consent to 90 days post last dose
Population: The safety population includes all participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 60 | 33 | 57
Participants
  Hyperbilirubinaemia | 0 | 2 | 1
  Hypercalcaemia | 1 | 0 | 0
  Hypercholesterolaemia | 1 | 0 | 1
  Hyperglycaemia | 4 | 2 | 1
  Hyperkalaemia | 2 | 1 | 2
  Hyperlipidaemia | 0 | 1 | 0
  Hypermagnesaemia | 1 | 0 | 0
  Hyperphosphataemia | 0 | 1 | 1
  Hypertriglyceridaemia | 1 | 0 | 0
  Hyperuricaemia | 3 | 5 | 2
  Hypoalbuminaemia | 2 | 0 | 2
  Hypocalcaemia | 3 | 1 | 1
  Hypokalaemia | 6 | 1 | 4
  Hypomagnesaemia | 2 | 2 | 1
  Hyponatraemia | 2 | 1 | 0
  Alanine Aminotransferase Increased | 1 | 0 | 3
  Aspartate Aminotransferase Increased | 1 | 0 | 3
  Blood Alkaline Phosphatase Increased | 1 | 1 | 2
  Blood Bilirubin Increased | 0 | 1 | 1
  Blood Cholesterol Decreased | 0 | 0 | 1
  Blood Creatinine Decreased | 1 | 0 | 0
  Blood Creatinine Increased | 1 | 2 | 1
  Blood Immunoglobulin G Decreased | 0 | 0 | 1
  Blood Lactate Dehydrogenase Increased | 4 | 0 | 0
  Blood Urea Increased | 1 | 1 | 0
  Gamma-Glutamyltransferase Increased | 1 | 1 | 2
  Hepatic enzyme Increased | 1 | 0 | 0
  Anaemia | 18 | 7 | 9
  Eosinophilia | 0 | 0 | 1
  Lymphopenia | 4 | 3 | 1
  Neutropenia | 28 | 10 | 19
  Thromobocytopenia | 12 | 6 | 10
  Activated Partial Thromboplastin Time Prolonged | 2 | 0 | 0
  Blood Fibrinogen Increased | 1 | 0 | 0
  Blood Immunoglobulin g Decreased | 0 | 0 | 1
  Haemoglobin Decreased | 0 | 1 | 0
  Lymphocyte Count Decreased | 3 | 0 | 2
  Neutrophil Count Decreased | 9 | 1 | 3
  Platelet Count Decreased | 2 | 2 | 3
  Prothrombin Time Shortened | 1 | 0 | 0
  Haematuria | 0 | 2 | 1
  Proteinuria | 0 | 1 | 0
  White Blood Cells in Urine | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Electrocardiogram Reported as AEs
Description: AEs observed in participants with clinically significant ECG abnormalities were assessed.
Time Frame: From time of consent to 90 days post last dose
Population: The safety population includes all participants who received any investigational product.
Measure: Number; unit: Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 60 | 33 | 57
Participants
  Atrial Fibrillation | 1 | 2 | 1
  Atrioventricular Block | 1 | 0 | 0
  Palpitations | 0 | 0 | 2
  Sinus Bradycardia | 1 | 0 | 0
  Sinus Tachycardia | 1 | 0 | 0
  Tachycardia | 2 | 1 | 1
  Pyrexia | 20 | 11 | 14
  Dyspnoea | 9 | 2 | 4
  Dyspnoea Exertional | 3 | 1 | 0
  Hypertension | 1 | 0 | 1
  Hypotension | 5 | 2 | 6
  Orthostatic Hypotension | 0 | 0 | 1

5. Secondary Outcome: Complete Response Rate
Description: Complete response was as per IWG was the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Percentage of Participants | 6.5 [1.8 to 15.7] | 5.6 [0.7 to 18.7] | 11.5 [4.7 to 22.2]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs MEDI-551 4 mg/kg + Bendamustine; Test type: Superiority or Other; p = 0.3206, Cochran-Mantel-Haenszel

6. Secondary Outcome: Minimal Residual Disease Negative Complete Response (CR) Rate
Description: The MRD-negative CR rate was defined as the percentage of participants who achieved CR and became MRD-negative as determined by flow cytometry. CR as per International Working Group (IWG) was complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Percentage of Participants | 1.6 [0.0 to 8.7] | 5.6 [0.7 to 18.7] | 4.9 [1.0 to 13.7]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs MEDI-551 4 mg/kg + Bendamustine; Test type: Superiority or Other; p = 0.3130, Cochran-Mantel-Haenszel

7. Secondary Outcome: Time to Response
Description: Time to response was evaluated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Months | 2.1 [1.9 to 2.6] | 1.9 [1.7 to 2.9] | 2.1 [1.9 to 3.5]

8. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined as the time from onset of treatment with study drug until first evidence/diagnosis of progressive disease or - in the absence of any diagnosis of progressive disease - until the participant´s death.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Months | 15.4 [12.0 to 27.2] | 15.0 [5.8 to 23.3] | 16.1 [12.5 to 24.0]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs MEDI-551 4 mg/kg + Bendamustine; Test type: Superiority or Other; p = 0.9527, Log Rank

9. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured from the start of treatment with study drug until the first documentation of disease progression or death due to any cause, whichever occurred first. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Months | 14.8 [11.4 to 23.5] | 15.0 [5.8 to 22.1] | 16.1 [12.5 to 21.6]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was determined as the time from the start of treatment with study drug until death due to any cause. For participants who were alive at the end of the study or lost to follow-up, OS was censored on the last date when the participant was known be alive. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population includes all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 62 | 36 | 61
Months | NA [NA to NA] — The median was not reached and the upper and lower limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — The median was not reached and the upper and lower limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [23.9 to NA] — The median was not reached and the upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

11. Secondary Outcome: Number of Participants Who Developed Detectable Anti-drug Antibodies (ADA)
Description: A participant was considered ADA-positive across the study if they had a positive reading at any time point during the study.
Time Frame: as for outcome 1
Population: The safety population includes all participants who received any investigational product. Participants whom ADA samples were available were analyzed for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 31 | 57
Participants | 4 | 8

12. Secondary Outcome: Terminal Half Life (t1/2) of MEDI-551
Description: Terminal phase elimination half-life (T1/2) was the time required for half of the drug to be eliminated from the serum.
Time Frame: Pre-infusion and 1 hour post infusion on Days 2 and 8, Days 15 and 22 of cycle 1
Population: The safety population includes all participants who received any investigational product. Participants whom PK samples were available were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Number analyzed (Participants) | 12 | 38
Day | 17.2 (9.56) | 22.0 (14.4)

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 90 days after the last dose of study drug
Arm/Group | Rituximab + Bendamustine | MEDI-551 2 mg/kg + Bendamustine | MEDI-551 4 mg/kg + Bendamustine
Serious Adverse Events (participants affected / at risk) | 19/60 | 16/33 | 19/57
Other Adverse Events (participants affected / at risk) | 58/60 | 31/33 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Bendamustine (N=60) | MEDI-551 2 mg/kg + Bendamustine (N=33) | MEDI-551 4 mg/kg + Bendamustine (N=57)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (3)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (5) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 5 (10) | 5 (14)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Bendamustine (N=60) | MEDI-551 2 mg/kg + Bendamustine (N=33) | MEDI-551 4 mg/kg + Bendamustine (N=57)
Anaemia (Blood and lymphatic system disorders) | 18 (64) | 7 (20) | 9 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (26) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (26) | 3 (7) | 1 (5)
Neutropenia (Blood and lymphatic system disorders) | 28 (78) | 10 (44) | 19 (58)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (76) | 5 (8) | 10 (21)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 3 (3) | 7 (15)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 20 (23) | 9 (11) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 13 (20) | 5 (5) | 11 (15)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (5)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 29 (45) | 13 (23) | 29 (47)
Vomiting (Gastrointestinal disorders) | 13 (14) | 7 (8) | 7 (7)
Asthenia (General disorders) | 20 (31) | 4 (4) | 7 (17)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 2 (2)
Chills (General disorders) | 11 (15) | 6 (7) | 7 (10)
Fatigue (General disorders) | 18 (38) | 14 (19) | 20 (30)
Oedema peripheral (General disorders) | 3 (4) | 2 (3) | 7 (7)
Peripheral swelling (General disorders) | 1 (2) | 1 (2) | 1 (2)
Pyrexia (General disorders) | 20 (27) | 11 (14) | 14 (23)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 1 (1) | 1 (2)
Bronchitis (Infections and infestations) | 4 (4) | 3 (4) | 4 (4)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (5) | 2 (3) | 4 (5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (8) | 0 (0) | 1 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 14 (25) | 21 (64) | 37 (123)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 0 (0) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 1 (2) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 2 (3) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 4 (7) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (4) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (8) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 9 (16) | 1 (3) | 3 (6)
Platelet count decreased (Investigations) | 2 (4) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 5 (6) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 13 (17) | 4 (4) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (6) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 1 (1) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 5 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (9) | 1 (1) | 7 (9)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5) | 3 (6) | 7 (10)
Dysgeusia (Nervous system disorders) | 5 (7) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 6 (9) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (2)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0) | 4 (5)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (7) | 2 (2) | 5 (5)
Dysuria (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 5 (9) | 19 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 2 (2) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (13) | 5 (9) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (7) | 4 (6) | 8 (10)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 4 (7) | 2 (3) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.